CLINICAL TRIAL: NCT06798038
Title: Comparison of the Efficacy of Chemical Genicular Nerve Neurolysis Using Alcohol or Phenol Versus Radiofrequency Ablation Under Ultrasound Guidance for Pain Management in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ghady Osama Makarem, Gomakarem, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36265MD337/12/24
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Assessment of Pain Intensity Using 10-point Numerical Rating Scale (NRS-10)(9)Immediately After Intervention , 1 Week,1month,3 Months,6months and One Year; Assessment of Knee Function Using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC); Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiofrequency Ablation; Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Radiofrequency ablation group (Experimental)
  Interventions: Device: radiofrequency ablation
- Alcohol injection group (Experimental)
  Interventions: Drug: alcohol neurolysis
- Phenol injection group (Experimental)
  Interventions: Drug: phenol neurolysis

INTERVENTIONS:
Device: radiofrequency ablation — 35 Patients will be undergo for radiofrequency ablation which will be applied to each genicular nerve.
  Arms: Radiofrequency ablation group
Drug: phenol neurolysis — 35 Patients will be administered with 2.0 ml of 6% phenol solution prepared from crystallized phenol per genicular nerve
  Arms: Phenol injection group
Drug: alcohol neurolysis — 35 Patients will be administered with 1.0ml of 70% alcohol per genicular nerve
  Arms: Alcohol injection group

SUMMARY:
Chronic knee pain is a common condition that affects many people, particularly those with knee osteoarthritis. It can limit mobility, reduce the quality of life, and increase the risk of falling .

There are various treatment options for chronic knee osteoarthritis pain, including medications, physical therapy and surgery. Topical and oral analgesic medications and physical therapy, are often used in this population but with variable success and often wanting pain relief over time as the condition progresses.

Patients who fail medical treatment often undergo total knee arthroplasty (TKA) However, there are significant comorbidities associated with TKA, and most of patients suffer with chronic knee pain after this surgery Furthermore, a subset of patients are unable to undergo TKA because of medical comorbidities.

One alternative treatment option is genicular nerve ablation, which involves destroying nerves that carry pain signals from the knee joint to the brain. Genicular nerve ablation can be performed using radiofrequency ablation (RFA) or chemical agents such as phenol. Both methods aim to provide long-term pain relief and functional improvement in patients with chronic knee pain(4).

Chemical neurolytics, such as alcohol or phenol, have come to the fore because of their low cost and ease of application compared to radiofrequency ablation.These methods can be easily applied with ultrasound (US) guidance, which allows precise targeting of the relevant nerves. However, there is a lack of literature on appropriate agents and dose selection issues .

Radiofrequency neurolysis (RFN) of the genicular nerves, which provides innervation to the capsule of the knee joint, as well as to the intra-articular and extra-articular ligaments, have been of considerable interest as an effective technique to alleviated knee osteoarthritis pain .However, it requires expensive specialized equipment and trained personnel, which may not be available or affordable in some settings.

ELIGIBILITY:
Inclusion Criteria:

* The following will be the criteria for inclusion, (105) patients older than 18 years with moderate to severe knee pain due to knee osteoarthritis (pain of intensity six or more on a numeric rating scale [NRS], persistent pain for more than six months, grade III or IV osteoarthritis in the radiological Kellgren-Lawrence (KL) classification (5-11), and failure to manage pain with conservative methods such as analgesics, intra-articular injection, and physical therapy.

Exclusion Criteria:

* • Patients' refusal to participate in the study.

  * History of intra-articular injection within three months before or after the procedure.
  * Coagulopathy and anticoagulant use.
  * Systemic disease as: renal or hepatic insufficiency.
  * Unable to communicate with the patient.
  * Implantable device.
  * Previous knee surgery.
  * Knee pain due to causes other than knee osteoarthritis (such as meniscopathy, trauma, spine disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity using 10-point numerical rating scale (NRS-10) | immediately after intervention , 1 week,1month,3 months,6months and one year.

SECONDARY OUTCOMES:
Assessment of Knee function using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | immediately after intervention , 1 week,1month,3 months,6months and one year.
2- Assessment of the side effects and complications of these methods as (paresthesia, motor deficits, pain during application and increase in pain) | immediately after intervention , 1 week,1month,3 months,6months and one year.